CLINICAL TRIAL: NCT03571672
Title: A Phase III, Open-Label, Multicenter Trial to Evaluate Ejection Fraction, End-Diastolic and End-Systolic Volumes, by Unenhanced and DEFINITY®-Enhanced 2D-Echo and Magnetic Resonance Imaging
Brief Title: DEF-314 Better Accuracy in Ejection Fraction (EF) Assessment With DEFINITY
Acronym: BENEFIT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DEF-314
Record Dates: First submitted 2018-06-06; First posted 2018-06-27 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Disease
Keywords: Left Ventricular Ejection Fraction; DEFINITY; Enhanced Echocardiogram; Cardiac Magnetic Resonance
MeSH Terms: conditions — Heart Diseases | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DEFINITY (Experimental): Each patient will undergo an unenhanced ultrasound examination and a DEFINITY contrast-enhanced ultrasound
  Interventions: Drug: DEFINITY

INTERVENTIONS:
Drug: DEFINITY — All subjects will receive a single dose of DEFINITY®

SUMMARY:
This is a Phase 3, prospective, open-label, multicenter study to evaluate Left Ventricular Ejection Fraction (LVEF) measurement accuracy and reproducibility of DEFINITY® contrast-enhanced and unenhanced echocardiography as compared with non-contrast cardiac magnetic resonance imaging (CMR) used as the truth standard.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age in sinus rhythm
2. Able to communicate effectively with trial personnel
3. Has undergone a 2D Echo with or without contrast obtained within 6 months prior to enrollment (Day 0)
4. Has provided signed informed consent after receiving a verbal and written explanation of this clinical trial -

Exclusion Criteria:

1. Female subjects who are pregnant or lactating. All women of child bearing potential [WOCBP] must have a negative urine pregnancy test at screening regardless of contraceptive use history.
2. Women of child-bearing potential are excluded unless they:

   1. are post-menopausal defined as amenorrhea ≥ 12 consecutive months, OR
   2. have undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy), OR
   3. have been using an adequate and medically approved method of contraception to avoid pregnancy for at least 1 month prior to DEFINITY® dose administration and be willing to continue using the same method for the duration of the study.
3. Current illness or pathology that would prevent undergoing investigational product administration due to a significant safety risk to the patient.
4. Uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 200 mmHg or diastolic blood pressure ≥ 110 mmHg) or arterial hypotension (defined as systolic blood pressure ≤ 90 mmHg).
5. Unstable cardiovascular status defined as:

   1. myocardial infarction or unstable angina pectoris within 6 months prior to enrollment/DEFINITY® dose administration day
   2. transient ischemic attack or stroke within 3 months prior to DEFINITY® dose administration
   3. symptomatic valvular heart disease or moderate to severe stenotic valvular heart disease
   4. clinically significant congenital heart defects
   5. current uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise
   6. acute pulmonary embolus or pulmonary infarction
   7. acute myocarditis or pericarditis
   8. acute aortic dissection
   9. atrial fibrillation
6. any major surgery within 4 weeks prior to screening
7. known contraindications to undergoing CMR or claustrophobia
8. participation in any investigational drug, device, or placebo study within 30 days prior to screening
9. known hypersensitivity to perflutren, or any of the excipients in DEFINITY®
10. prisoners or those who are subject to compulsory detention or involuntary incarceration for treatment of either a psychiatric or physical illness (e.g., infectious disease) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of California-San Diego, San Diego, California
  - Alfieri Cardiology, Wilmington, Delaware
  - Henry Ford Hospital, Detroit, Michigan
  - Weill Cornell Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospital/Cleveland Medical Center, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Virginia University Medical Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Definity
Started | 153
Completed | 148
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Baseline data are calculated based on Safety Population
Arm/Group | Definity
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 98
  >=65 years | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 135
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 37
  White | 104
  More than one race | 3
  Unknown or Not Reported | 0
LVEF Group [Count of Participants; unit: Participants] — Left Ventricular Ejection Fraction (LVEF) Percentage measured by Cardiac Magnetic Resonance (CMR) imaging
  Participants
    LVEF <30% | 35
    LVEF 30-40% | 40
    LVEF 41-50% | 39
    LVEF >50% | 39

OUTCOME MEASURES:

1. Primary Outcome: Absolute Value of LVEF Percentage Differences From CMR by Blinded Reader
Description: Demonstrate improvement in accuracy in left ventricular ejection fraction (LVEF) assessment using Definity contrast-enhanced over unenhanced echocardiography by comparing LVEF Percentage Differences from CMR measured by 3 independent blinded image readers.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Groups:
- Blinded Reader 1: Independent Blinded Reader 1 of 3
- Blinded Reader 2: Independent Blinded Reader 2 of 3
- Blinded Reader 3: Independent Blinded Reader 3 of 3
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 145 | 145 | 145
Percent Ejection Fraction
  Echo Enhanced | 6.10 (5.319) | 6.38 (5.227) | 4.93 (4.288)
  Echo Unenhanced | 6.18 (5.300) | 6.61 (5.256) | 5.36 (4.498)
Statistical Analysis 1: Comparison: Blinded Reader 1; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.868, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.08, Standard Deviation 5.980
Statistical Analysis 2: Comparison: Blinded Reader 2; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.606, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.23, Standard Deviation 5.445
Statistical Analysis 3: Comparison: Blinded Reader 3; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.224, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.43, Standard Deviation 4.212

2. Secondary Outcome: Secondary Objective 1: Absolute Value of LVEF Percentage Differences From CMR by Blinded Reader for Suboptimal Echocardiograms
Description: Demonstrate improvement in accuracy in left ventricular ejection fraction (LVEF) assessment using DEFINITY® contrast-enhanced over unenhanced echocardiography in subjects with suboptimal echocardiograms by comparing LVEF percentage differences from CMR measured by 3 independent readers.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Per-protocol population - Sub-optimal Echocardiograms
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 59 | 59 | 59
Percent Ejection Fraction
  Echo Enhanced | 7.48 (6.228) | 7.16 (6.337) | 5.71 (5.293)
  Echo Unenhanced | 7.16 (6.184) | 7.12 (5.381) | 5.89 (4.523)
Statistical Analysis 1: Comparison: Blinded Reader 1; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.715, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.32, Standard Deviation 6.682
Statistical Analysis 2: Comparison: Blinded Reader 2; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.956, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.05, Standard Deviation 6.526
Statistical Analysis 3: Comparison: Blinded Reader 3; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.771, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.17, Standard Deviation 4.584

3. Secondary Outcome: Secondary Objective 2: Absolute Value LVEF Percentage Differences From CMR Between Blinded Readers
Description: Demonstrate a reduction in inter-reader variability for the assessment of left ventricular ejection fraction using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing LVEF Percentage Differences from CMR between 3 independent blinded readers
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 145 | 145 | 145
Percent Ejection Fraction
  Echo Enhanced | 6.10 (5.319) | 6.38 (5.227) | 4.93 (4.288)
  Echo Unenhanced | 6.18 (0.164) | 6.61 (5.256) | 5.36 (4.498)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.959, 95% CI 2-sided [0.944 to 0.970]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.950, 95% CI 2-sided [0.931 to 0.964]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.957, 95% CI 2-sided [0.941 to 0.969]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.934, 95% CI 2-sided [0.909 to 0.952]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.961, 95% CI 2-sided [0.946 to 0.972]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.937, 95% CI 2-sided [0.913 to 0.954]

4. Secondary Outcome: Secondary Objective 3: Absolute Value End-Diastolic and Systolic Volume Differences From CMR Between Blinded Readers
Description: Demonstrate a reduction in inter-reader variability for the assessment of end-diastolic and systolic volumes using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing end-diastolic and systolic volume differences from CMR between 3 independent blinded readers.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 145 | 145 | 145
mL
  Echo Enhanced End Diastolic | 52.31 (35.726) | 46.57 (33.785) | 39.37 (26.206)
  Echo Unenhanced End Diastolic | 58.02 (38.483) | 56.65 (37.766) | 48.07 (31.620)
  Echo Enhanced End Systolic | 33.56 (28.641) | 29.93 (25.845) | 26.01 (20.740)
  Echo Unenhanced End Systolic | 37.53 (30.016) | 33.51 (28.079) | 30.72 (23.534)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.988, 95% CI 2-sided [0.984 to 0.992]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.986, 95% CI 2-sided [0.981 to 0.990]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.960, 95% CI 2-sided [0.945 to 0.971]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.925, 95% CI 2-sided [0.897 to 0.945]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.970, 95% CI 2-sided [0.958 to 0.978]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.909, 95% CI 2-sided [0.876 to 0.934]
Statistical Analysis 7: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.989, 95% CI 2-sided [0.984 to 0.992]
Statistical Analysis 8: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.985, 95% CI 2-sided [0.979 to 0.989]
Statistical Analysis 9: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.973, 95% CI 2-sided [0.962 to 0.980]
Statistical Analysis 10: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.947, 95% CI 2-sided [0.927 to 0.961]
Statistical Analysis 11: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.977, 95% CI 2-sided [0.969 to 0.984]
Statistical Analysis 12: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.937, 95% CI 2-sided [0.914 to 0.954]

5. Secondary Outcome: Secondary Objective 4: Absolute Value of LVEF Percentage Differences From CMR Between Blinded Readers for Suboptimal Echocardiograms
Description: Demonstrate a reduction in inter-reader variability for the assessment of left ventricular ejection fraction using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing LVEF Percentage Differences from CMR between 3 independent blinded readers in subjects with suboptimal echocardiograms.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Per Protocol Population - Sub-Optimal Echocardiograms
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 59 | 59 | 59
Percent Ejection Fraction
  Echo Enhanced | 7.48 (6.228) | 7.16 (6.337) | 5.71 (5.293)
  Echo Unenhanced | 7.16 (6.184) | 7.12 (5.381) | 5.89 (4.523)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.945, 95% CI 2-sided [0.909 to 0.967]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.917, 95% CI 2-sided [0.864 to 0.950]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.939, 95% CI 2-sided [0.900 to 0.963]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.894, 95% CI 2-sided [0.827 to 0.935]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.952, 95% CI 2-sided [0.920 to 0.971]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.900, 95% CI 2-sided [0.838 to 0.939]

6. Secondary Outcome: Secondary Objective 5: Absolute Value End-Diastolic and Systolic Volume Differences From CMR Between Blinded Readers for Suboptimal Echocardiograms
Description: Demonstrate a reduction in inter-reader variability for the assessment of end-diastolic/systolic volumes using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing end-diastolic and systolic volume differences from CMR between 3 independent blinded readers in subjects with suboptimal echocardiograms.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT population - Sub Optimal Echocardiograms
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 59 | 59 | 59
mL
  Echo Enhanced End Diastolic | 62.34 (40.035) | 54.68 (37.571) | 45.44 (29.702)
  Echo Unenhanced End Diastolic | 65.45 (43.227) | 63.25 (41.700) | 53.77 (34.210)
  Echo Enhanced End Systolic | 39.52 (29.712) | 34.00 (26.955) | 30.12 (22.174)
  Echo Unenhanced End Systolic | 39.45 (33.303) | 33.97 (29.233) | 32.78 (24.522)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.976, 95% CI 2-sided [0.961 to 0.986]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.984, 95% CI 2-sided [0.974 to 0.991]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.933, 95% CI 2-sided [0.890 to 0.960]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.857, 95% CI 2-sided [0.770 to 0.912]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.948, 95% CI 2-sided [0.914 to 0.969]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.824, 95% CI 2-sided [0.721 to 0.892]
Statistical Analysis 7: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.982, 95% CI 2-sided [0.970 to 0.989]
Statistical Analysis 8: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.974, 95% CI 2-sided [0.957 to 0.985]
Statistical Analysis 9: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.948, 95% CI 2-sided [0.915 to 0.969]
Statistical Analysis 10: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.890, 95% CI 2-sided [0.822 to 0.933]
Statistical Analysis 11: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.959, 95% CI 2-sided [0.932 to 0.975]
Statistical Analysis 12: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.872, 95% CI 2-sided [0.794 to 0.922]

ADVERSE EVENTS:
Time Frame: Up to 12 days: Enrolled subjects were followed for adverse events and serious adverse events from the time the Informed Consent was signed at screening (Day -7 to Day 0) through 72+/- 24 hours after completion of Definity administration (Day 0).
Groups:
- Definity: Each patient will undergo an unenhanced ultrasound examination and a single dose DEFINITY contrast-enhanced ultrasound during the same imaging session
Arm/Group | Definity
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 0/153
Other Adverse Events (participants affected / at risk) | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03571672/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03571672/SAP_001.pdf